CLINICAL TRIAL: NCT05306691
Title: Comparative Remineralizing Efficacy of Giomer Bioactive Barrier Varnish vs. Fluoride Varnish in Management of White Spot Lesions in Adult Patients: Randomized Controlled Tria
Brief Title: Remineralizing Efficacy of Giomer Varnish vs. Fluoride Varnish in Management of White Spot Lesions in Adult Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Amr Mohamed Kotb, Master degree student, Conservative Dentistry Department Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Giomer Bioative varnish
Record Dates: First submitted 2022-03-02; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Caries, Dental; Remineralization; White Spot Lesion
MeSH Terms: conditions — Dental Caries | interventions — PRG Barrier Coat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bio-smart Light Cured Protective Shield with bioactive S-PRG filler technology (PRG Barrier Coat) (Experimental): Surface reaction-type pre-released glass ionomer (S-PRG) fillers containing dental materials are now commercially available. It was shown that PRG filler is an active ingredient with the ability to release and recharge fluoride ions. In addition, S-PRG fillers release five other active ions, Sr2þ, SiO3 2, Naþ, BO3 3, and Al3þ. S-PRG filler has a modulation effect on acidic conditions, causing the surrounding environment to become weakly alkaline upon contact with water or acidic solutions. This effect was thought to be brought by Sr, B, Na, and F ions released from S-PRG filler. A fluoride-releasing coating material containing S-PRG filler (PRG BarrierCoat®, SHOFU, Japan) was manufactured as a coating material to suppress dentin hypersensitivity and prevent caries on smooth surface areas
  Interventions: Drug: Bio-smart Light Cured Protective Shield with bioactive S-PRG (Surface Pre- Reacted Glass ionomer) filler technology (PRG Barrier Coat) by (By SHOFU Inc., Japan).
- 5% NaF varnish (Proflourid Varnish VOCO America Inc.). (Active Comparator): The gold standard remineralizing agent recommended by the guidelines
  Interventions: Drug: Bio-smart Light Cured Protective Shield with bioactive S-PRG (Surface Pre- Reacted Glass ionomer) filler technology (PRG Barrier Coat) by (By SHOFU Inc., Japan).

INTERVENTIONS:
Drug: Bio-smart Light Cured Protective Shield with bioactive S-PRG (Surface Pre- Reacted Glass ionomer) filler technology (PRG Barrier Coat) by (By SHOFU Inc., Japan). — Surface reaction-type pre-released glass ionomer (S-PRG) fillers containing dental materials are now commercially available. It was shown that PRG filler is an active ingredient with the ability to release and recharge fluoride ions. In addition, S-PRG fillers release five other active ions, Sr2þ, SiO3 2, Naþ, BO3 3, and Al3þ. S-PRG filler has a modulation effect on acidic conditions, causing the surrounding environment to become weakly alkaline upon contact with water or acidic solutions. This effect was thought to be brought by Sr, B, Na, and F ions released from S-PRG filler. A fluoride-releasing coating material containing S-PRG filler (PRG BarrierCoat®, SHOFU, Japan) was manufactured as a coating material to suppress dentin hypersensitivity and prevent caries on smooth surface areas.

SUMMARY:
To evaluate the remineralizing capability of biosmart S-PRG barrier coat varnish and its employment in clinical practice

ELIGIBILITY:
Inclusion Criteria:

* • Age range between 18 and 40 years.

  * Patients with no systemic diseases, syndromic abnormalities, or proven/suspected milk protein allergy and/or sensitivity
  * Patients with fair oral hygiene (mild to moderate plaque accumulation).
  * Patients with non-cavitated initial carious lesions grade 0 or 1 caries in accordance with The Nyvad caries diagnostic criteria.
  * The patient did not receive any remineralizing agent other than the regular toothpaste during the past three months.

Exclusion Criteria:

* • Severe or active periodontal disease.

  * Patients had received therapeutic irradiation to the head and neck region.
  * Patients had participated in a clinical trial within 6 months before commencement of this trial.
  * Patients unable to return for recall appointments
  * Presence of abnormal oral, medical, or mental condition.
  * Presence of dentin caries or enamel hypoplasia on maxillary anterior teeth.
  * Patients with glass ionomer restorations because the glass ionomer restoration release fluoride in the oral cavity, potentially impacting the results.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Remineralization efficacy. | Baseline, 1 month, 3 months
  Determination of lesion level by DIAGNOdent which provides a laser fluorescence feedback to give a numerical readout reflecting the amount of demineralization

SECONDARY OUTCOMES:
Change in Caries lesion activity assessment | Baseline, 1 month, 3 months
  Visual- tactile. The Nyvad criteria is a visual-tactile caries classification system designed to detect the activity and severity of caries lesions, the diagnostic criteria reflect the entire continuum of caries, ranging from clinically sound surfaces to non-cavitated and microcavitated caries lesions in enamel to frank cavitation into the dentine